**Study Title:** RealConsent: A web-based program to reduce college women's risk of sexual violence by targeting alcohol use, communication and consent, and building supportive networks.

**Date of Document**: July 31, 2018

# Georgia State University Department of Health Promotion and Behavior School of Public Health

#### **Research Protocol and Statistical Analyses**

Title: Testing the efficacy of a web-based program for college women

Principal Investigator: Dr. Laura F. Salazar

Sponsor: National Institute of Alcohol Abuse and Alcoholism

### I. Project Summary and Project Goals

Sexual assault of college women is a serious and complex public health problem: one in five college women report being sexually assaulted. The purpose of this study is to conduct a randomized controlled trial study with 750 female college students from three universities to test the efficacy of RealConsent-F, a sexual violence risk reduction program for college women, compared to an attention-placebo comparison condition. The primary outcome will be self-reported sexual violence victimization and the secondary outcomes will be alcohol and dating protective- and risk-related behaviors and resistance strategies. Our expected outcomes are demonstrated feasibility and efficacy of a technologically novel risk reduction program for female college students.

## II. Rationale and Background Information

Epidemic of Sexual Violence Against College Women: Recent statistics on sexual violence against women in college have revealed a serious and complex public health problem: 6% of female college students report experiences of rape each year<sup>14</sup> and one in five women report that she was sexually assaulted while in college. Assaults typically occur during freshman or sophomore year<sup>2</sup> and, in most cases (75-80%), women state that they know their attacker, whether as an acquaintance, classmate, friend or (ex)boyfriend. Many women report experiencing an "incapacitated assault" meaning they were sexually abused while they, the victims, were drugged, drunk, passed out, or otherwise incapacitated. These data demonstrate the high level of sexual assault occurring among young adult college women. To reduce incidence rates, comprehensive approaches involving evidence-based, easily-disseminated educational products are greatly needed by institutions of higher learning to prevent male perpetration and reduce risk of sexual assault among women; however, evidence-based prevention and risk reduction programming is greatly lacking. For

In 2014 the Centers for Disease Control and Prevention (CDC) conducted a review of 140 published sexual violence primary prevention interventions and concluded *only three* were

effective in <u>preventing</u> sexual violence perpetration. [Note: RealConsent male version (RealConsent-M) was not included in this review as the publication was "in press" at the time the review was conducted]. Of the three effective programs, <u>none</u> were specific to college students. To <u>reduce sexual violence perpetration</u>, best practices for prevention entail theoretically-driven activities that focus on improving 1) knowledge of consent and understanding the impact of alcohol; 2) addressing hyper-male ideology; 3) reducing hostility toward women; 4) reducing adherence to prescribed gender roles; 5) changing social norms to reduce acceptance of sexual violence; 6) dispelling rape myths; and 7) enhancing communication skills between men and women around sex. RealConsent-M incorporated segments that addressed all seven best practices. Using a randomized controlled trial (RCT), RealConsent-M demonstrated significant reductions in sexual violence perpetration; thus, RealConsent is the first effective prevention program for male college students.

#### III. Methods

This study plans to conduct a randomized controlled trial with 750 female freshmen between 18-20 years of age from three universities in the state of Georgia (n=250 from each school) to test the efficacy of RealConsent-F compared to an attention-placebo comparison condition. Inclusion criteria for all proposed research activities are: female, aged 18-20 years, full time freshman, and single. Exclusion criteria are: other education levels, married, and/or graduate status. Participants will be randomized to either the intervention or attention-placebo study conditions. To control for Hawthorne effects, women in the RCT will be compared to women in an attention-placebo control condition—a general health promotion web-based program called "Stress Management." Below are descriptions of the intervention, RealConsent and the attention-placebo program.

#### RealConsent-F

RealConsent includes 18 of 40 well-known behavioral change techniques. The program 1) provides <u>information</u> on the targeted behavior; 2) provides <u>instruction</u> on how to perform the behavior; 3) demonstrates or <u>models</u> the behavior; 4) demonstrates <u>positive outcomes</u> for engaging in the behavior or <u>negative outcomes</u> for failing to change behavior; and 5) provides encouragement and positive feedback as <u>reinforcement</u>. RealConsent-F uses didactic methods involving presentation of material via video; problem-based learning via quizzes with interactivity; short videos and animation to model the behavior. RealConsent-F is unique in that it includes serial drama episodes (i.e. "Squad") featuring four college women going through their freshman year and experiencing issues related to alcohol use, sexual assault, stalking, and dating violence. This program is grounded in *educational entertainment* to provide educational content within entertainment programming (e.g., Sesame Street or Law and Order).

# Attention-Placebo Condition

Stress Management was developed by ISA Group (www.isagroup.com) and is a multi-media web-based program designed to help manage stress levels. The program is dynamic and interactive with substantial use of video/audio. Each of 4 program modules is ≈30 minutes involving interactive and didactic activities. Thus, it approximates RealConsent-F in format and duration.

#### Recruitment of N=750 Female College Freshmen

We have agreements with each of the three colleges to test RealConsent-F among female freshmen and they have agreed to provide a list of female students. We will send out email invites from Salazar's email account to a random sample of 500 students per school to ask for their participation in a research project. To control for demand characteristics, we will blind participants to the research question and indicate the purpose is to "test multimedia, web-based interactive programs designed for female college students." If the first round of 500 emails does not produce a 50% response rate, we will send out another batch of 500 email invites to reach our target goal of n=250 at each college. Salazar used this recruitment strategy for testing RealConsent-M. Female freshmen who are interested in the research will be able to access our online eligibility screener through a hyperlink in the body of the email that takes them to our study website. Mr. Long, a computer scientist and programmer, will develop the study website and a web-based application that will help our project director with recruitment and retention efforts. Long developed a website and app for Salazar's current online study of 1,800 male freshmen.

#### Informed Consent

The website will provide a short description of the study and, if interested, participants can click on a button to assess their eligibility followed by the informed consent process. The informed consent process is a crucial aspect of any study, but especially so when conducting web-based research involving sensitive topics. Special consideration must be made to ensure that participants are aware of their rights as participants in such research. A hyperlink will be displayed following the eligibility screener directing eligible participants to the informed consent form. Those not eligible will receive a message saying they are not eligible. An interactive process will be designed to secure informed consent. As part of registration, we will collect name, preferred email, mailing address, and cell phone number to maximize retention although identifying information will not be linked with survey data. The web app will allow us to collect key data for CONSORT. All participants are eligible to receive up \$105 in Amazon e-gift cards for completing RealConsent-F and all surveys, which in our experience of 10 years of conducting online studies is feasible and necessary. \$13,96-98

# Baseline Assessment, Randomization, and Completion of RealConsent or Stress Management:

Once a participant is registered, she will get a confirmation email; her response will trigger another email that contains a link to the online baseline survey and a password for accessing. To enhance confidentiality of responses, we will encourage participants to choose a private location, use a secure, encrypted Internet connection, and close their web-browser after they have completed a survey. Once an individual completes the baseline survey, she will be randomized using an automated stratified block randomization program to either RealConsent-F or to Stress Management programs. Stratified block randomization will ensure equal numbers between conditions and that 125 participants from each university are assigned to each condition.

We will communicate to the research participants and encourage them to complete their assigned task (RealConsent-F or Stress Management) within two weeks. Participants can complete the modules at their own pace within the 2-week window and are able to leave a module and finish it later. Email prompts will be sent every 48 hours to remind participants to complete the modules. Participants will be contacted by email and/or text message prior to 6 months post-intervention (Spring 2019) to complete the posttest.

#### **Retention Activities**

Based on the experience and expertise of Salazar and her team, we will employ a number of activities to maximize retention. In a preliminary study of N=1,153 college male freshmen assessed three times over 12 months, Salazar and colleagues implemented activities to enhance recruitment: 1) sending touch-point emails in between assessments; 2) enabling participants to update changes in contact information via the web application; 3) providing full incentive amount for those who completed assessments on time as a "bonus;" 4) sending email and text reminders prior to due dates; and 5) emailing, texting and making phone calls up until final date. Our response rates were: 80% at wave 2 (6-months), and 81% at wave 3 (12-months). To ensure we maintain at least 80% retention rate, we will employ these strategies and those used previously by Salazar in other studies involving follow-up assessments of adolescents and adults.

#### Study Measures

The table below displays the measures that will be used in all study assessments.

**Table 1. Measures of Study Variables** 

| Variable | Measure | # Items | α |
|---|---|---|---|
| Primary Outcome:<br>Sexual Victimization | Revised Sexual Experiences Survey-SFV (SES) <sup>8</sup> | 35 | .74 |
| Secondary Outcomes: Dating behaviors | The Dating Behavior Survey (DBS) <sup>82,83</sup> | 15 | .67 |

| | The Dating Self-Protection Against Rape Scale <sup>83,84</sup> | 15 | .88 |
|---|---|---|---|
| Alcohol Protective Behaviors | Protective Behavioral Strategies Survey <sup>26,85</sup> | 15 | .94 |
| Use of resistance tactics | Use of Resistance Tactics <sup>23</sup> | 6 | n/a |
| Mediators: | | | |
| Alcohol use | Weekly Drinking and Heavy Episodic Drinking <sup>28,86</sup> | 2 | n/a |
| Perceptions of Alcohol-Related Risk | Likelihood of nonconsensual sex due to alcohol <sup>87</sup> | 1 | n/a |
| Alcohol Expectancy | Revised Alcohol Expectancy Questionnaire 87,888 | 40 | .72 |
| Alcohol Use Norms | Drinking norms rating form <sup>26,89</sup> | 1 | n/a |
| Bystander Behavior | Bystander Behavior Scale | 10 | .89 |
| Knowledge of legal definitions of rape | Legal Knowledge Scale <sup>13</sup> | 7 | .69 |
| Perceptions of informed consent | Informed Consent Index <sup>13</sup> | 14 | n/a |
| Empathy for rape victims | Rape Empathy Scale <sup>90</sup> | 19 | .84 |
| Communication with partner about sex | Communication subscale of SSBQ <sup>91</sup> | 7 | .80 |
| Sexual Assertiveness | Sexual Communication Survey <sup>82</sup> | 10 | .90 |
| Self-efficacy to discuss sex | Communication Self-Efficacy <sup>92</sup> | 4 | .84 |
| Self-efficacy to use assertive responses | Self Efficacy Scale <sup>93</sup> | 7 | .97 |
| Use of risk reduction strategies | Personal and Social Risk Reduction Strategies Scale | 34 | n/ŧ |

#### IV. Safety Considerations

There are some potential risks for participating in the RealConsent program. Participants may experience some adverse psychological reactions such as feeling upset or discomfort as they undergo the intervention modules. For example, a potential risk is that a participant may gain a new awareness of an unwanted sexual experience that hitherto she thought of as "her fault for getting drunk", but she now may indicate she was a victim of date rape. Although these instances represent some degree of risk, we have designed the procedures to minimize adverse reactions. Our project director, Dr. Anne Marie Schipani-McLaughlin will conduct a check-in with each participant after completion of each intervention module. Participants can freely elect to terminate participation in the Web-based intervention if so desired. We anticipate that some participants may require counseling and we will be prepared to help these participants with appropriate referrals. Dr. Schipani-McLaughlin has extensive experience in addressing participants' concerns during randomized trials will also undergo training by Dr. Salazar and if needed, the principal investigator will address adverse reactions should they arise. Also, we will include on our study website a (800 715 4225) number that can be accessed 24/7 for immediate crisis counseling in GA (GA Crisis and Access Line):

http://www.armstrong.edu/Departments/counseling\_center/counseling\_georgia\_crisis\_and\_access\_line).

Another potential risk for participating is the administered assessments that may cause some participants to experience adverse psychological reaction such as distress, discomfort, or anxiety responding to explicit questions regarding their unwanted sexual experiences. We will state explicitly that participants can refuse to answer any questions, decline to answer any questions, or be allowed to skip any questions of the survey; they can also elect to terminate their participation immediately. The project director will be prepared to provide resources for participants should they request a referral, or as they respond to explicit questions regarding their unwanted sexual experiences.

One last risk entails a loss of confidentiality. A number of steps will be taken to secure sensitive data. These include the required use of personal identification numbers, access codes, and passwords on the study web site and on all web-administered surveys and assessments. Only the PI and the project director will have access to the online survey data through our Qualtrics account. Qualtrics web-survey platform employs a high level of data encryption. We will also secure the web site, which will deliver the RealConsent program. All data and recruitment materials will be stored on the PI's password-protected desktop located in her locked office at GSU.

# V. Data Management and Statistical Analysis

#### Data Management

Data will be stored on servers that are protected by high-end firewall systems, data are encrypted so that information cannot be decoded, and IP addresses will not be collected (every computer that communicates over the Internet is assigned an IP address that uniquely identifies the device). Data files, once downloaded, will be stored on Dr. Salazar's password-protected computer located in her locked office.

#### Statistical Analysis

The complex empirical methods described below will be conducted by Dr. Hayat, an experienced statistician and colleague of Dr. Salazar's. Data analysis will be performed using the SAS Software System. Descriptive statistics for all measurements will be estimated and reported. Frequency distributions will be created to screen for any errors and will be used to summarize categorical data; measures of central tendency and dispersion will be used to summarize continuous data. All data will be examined for bivariate relationships and results used to build a multivariate statistical model.

We will analyze our study data with an intent-to-treat and per protocol analyses. An intent-to-treat analysis includes all participants who were randomized, regardless of compliance, withdrawal, and anything that happens after randomization. An advantage is that it is an analysis based on original randomization; however, effect estimation may be conservative and misleading with increasing attrition. A per protocol analysis considers only participants who fully complied and completed the study. Per protocol is less conservative and may reflect true treatment differences for those with full compliance. Including an intent-to-treat and per protocol analysis will provide a more complete understanding of treatment effects. Because we will most likely encounter incomplete data due to dropouts and non-response, multiple imputation of missing data will be used to impute missing values based on other available covariates.

Outcomes, including victimization and frequency of risky dating behaviors and alcohol-protective behaviors will be modeled using a general linear mixed model. This is an appropriate statistical model to use with repeated measures data collected over time. A random effect for subject will be included to account for the multiple measurements taken at baseline and 6-month follow-up on each subject. Treatment group and demographics will be included as fixed effects in the model. Mediation models will be tested with a two-tiered approach for mediation testing, with bootstrapping to generate estimates of the indirect effect and 95% confidence intervals.

#### Sample Size

Primary outcome will be report of victimization; secondary outcomes are protective- and risk- related behaviors. Sample size is based on the number per group needed to detect clinically meaningful treatment effects on victimization. Calculations were based on 80% power, level of significance of .05, and two- tailed statistical tests. Clinically meaningful treatment efficacy was defined for our outcome variable as having between a small and moderate effect size (Cohen's  $h \ge .35$ ). This effect size was considered as a 9% point difference between groups, at a minimum, and could potentially translate to a clinically significant reduction in the number of victimizations on those college campuses that implement RealConsent. Based on previous research with female college students,  $^{22,23,26,28,104-107}$  assuming incidence of 0.22 without intervention and .13 with intervention, a total of 558 participants are needed (279 in each group). We expect 20% attrition based on previous work. To achieve adequate power, we estimate a needed sample size of at least 670; however, we are increasing sample size to 750 participants (375 in each group) to increase power.

#### VI. Quality Assurance

# Data Safety & Monitoring Plan

In accordance with the NIH recommendations as this is a NIH clinical trial we will have a Data Safety Monitoring Board (DSMB). The proposed study is considered to present minimal risk to participants, given that they will complete surveys and possibly participate in a sexual violence prevention educational program. Members of the DSMB will perform the following activities:

- 1. Review the research protocol and plans for data and safety monitoring.
- 2. Review progress of the trial, including analysis of data quality and timeliness; subject recruitment and retention; subject risk versus benefit; and other factors that may affect outcome.
- 3. Review serious adverse event reports, provide commentary, and provide oversight to ensure that reports are relayed to individual IRBs and to the Office of Human Research Protections (OHRP), as indicated.
- 4. Review analyses of outcome data and review reports of related studies to

- determine whether the current study needs to be changed or terminated.
- 5. Determine whether the trial should continue as designed, should be changed, or should be terminated based on the data and make recommendations to the NIH and the Institutional Review Board considering conclusion or continuation of the study.
- 6. Review proposed modifications to the study prior to their implementation.
- 7. Protect the confidentiality of the trial data and the results of the monitoring.
- 8. Determine whether and to whom outcome results should be released prior to the reporting of study results.
- 9. Following DSMB meetings, provide appropriate NIH staff with written information concerning their findings.

The DSMB members will be chosen by Dr. Salazar and will be reviewed and approved by the NIH Project Officer. The members, who will all be voting members, will be chosen based upon their knowledge of clinical trial methodology, their experience with the topical area (i.e., sexual violence risk reduction strategies), and absence of conflicts of interest. They will be appointed for the life of the project. The Chair of the DSMB will be selected from among the DSMB members. The NIH Project Officer will serve as an ex-officio member of the DSMB.

DSMB meetings will be held every 12 months beginning in Year 1 of the study. Serious adverse events will be reported to the Chair as soon as they occur. The Chair of the DSMB will determine whether an in-person meeting or teleconference is needed. Prior to the meetings, a written report containing any study preliminary findings will be sent to DSMB members. Preliminary findings will not be made available to individuals outside of the DSMB. Each meeting will include time to review the progress of the study and to answer questions from members of the DSMB. Members of the DSMB will disclose any potential conflicts of interest, either pre- existing or those that develop during their tenure, to the Principal Investigator and the NIH Project Officer.

In accordance with NIH policy, a data and safety monitoring plan has been developed for the proposed study. Dr. Salazar will provide oversight of all recruitment and study procedures and quality assurance checks will be conducted as planned. All records pertaining to the study and all of the original and electronic files containing collected data will be securely stored. Dr. Salazar and will be solely responsible for dissemination of study findings through presentation and publication formats. Presentations and publications will not disclose the name of the clinics where recruitment occurred. Dr. Salazar will also be solely responsible for handling any requests from other investigators to examine the data collected during Phase II of this Fast- track proposal. Dr. Salazar will present these requests to a Data and Safety Monitoring Board (DSMB) for their consideration.

This research team has extensive experience working with college student populations and extensive experience confronting ethical issues of subjects in behavioral

interventions. We will work with all respective IRBs involved to assure compliance with ethical and HIPPA standards. Additionally, no incentives (i.e., "finder's fees) will be provided to staff for recruiting or referring subjects into the study. Moreover, we are going to make it abundantly clear to subjects that participation in the study will in no way affects their standing at their academic institutions.

Procedures for Monitoring Adverse Events. All study personnel, will be trained regarding how to handle adverse events. Possible adverse events that are unanticipated will be brought to the attention of the PIs, the IRBs, and the NIH project officer. The IRBs who will determine whether it is appropriate to stop the study protocol temporarily or will provide suggestions/modifications to the study procedures as necessary. Possible modifications include adding these possible adverse events to the consent form and reconsenting all study subjects. The PIs will be responsible for monitoring participant safety on a monthly basis at regularly scheduled research meetings. They will keep a written log of all events and ensure that the IRBs are contacted immediately. They will also keep a log of the outcome of IRB decisions regarding adverse events and apprise the research team of any changes that need to occur as a result of IRB decisions.

- 1. Dr. Salazar will provide oversight of all recruitment and study procedures and quality assurance checks will be conducted by the Project Director Dr. Schipani-McLaughlin as planned. These quality assurance checks will occur once a week during recruitment and assessment time periods to ensure recruitment goals and validity of the data.
- 2. All records pertaining to the study and all of the original and electronic files containing collected data will be securely stored by Dr. Salazar on her password-protected desktop computer and/or a locked file cabinet located in her locked office on GSU campus. Other than Dr. Salazar, only key study personnel will have access to the data files.
- 3. Specific procedures to ensure the safety of participants will also occur. The proposed research contains some risk for participants; however, the likelihood of adverse events (AEs) is low. During the efficacy trial, we will contact participants via email and texting to not only check in with them but also to promote compliance. All participants who demonstrate they are in need of assistance will be given a 800 telephone number to obtain immediate crisis counseling and a referral 24/7; thus, young women will have access to help in the event they feel distress or are upset.
- 4. Dr. Salazar will participate in the monitoring of participants during the course of the research. Should any AEs occur, the project director will be required to immediately contact Dr. Salazar. Dr. Salazar will immediately investigate the event and determine the appropriate manner in which to proceed. A report describing the AE will be submitted to the participating Institutional Review Board and to the project officer from NICHD within 10 days of occurrence. In the event a change in procedures is required, an amendment to IRB will occur

- promptly, within 10 days.
- 5. To monitor that our recruitment and retention projections are being met, Dr. Salazar will hold weekly meetings of the research team to assess recruitment and retention of participants.
- 6. Drs. Salazar and Hayat will be responsible for dissemination of study findings through presentation and publication formats. The setting for this research will not be named in publications or presentations.
- 7. Dr. Schipani-McLaughlin, the project director will monitor the data on a weekly basis during assessment periods. She will serve as the project data manager where she will examine the data for accuracy and any inconsistencies. She will rectify any errors and she will maintain a data correction log to record any errors and how they were resolved.
- 8. Dr. Matt Hayat, a Co-investigator and statistician on the study, will also perform interim analyses to assess the integrity of the data.
- 9. Finally, Dr. Salazar, will monitor the study using the following criteria:
  - a) Review progress of the surveys as they occur, including analysis of data quality and timeliness; subject recruitment, and other factors that may affect outcome.
  - b) Review serious adverse event reports, provide commentary, and provide oversight to ensure that reports are relayed to individual IRBs and to the Office of Human Research Protections (OHRP), as indicated.
  - c) Review analyses of outcome data of the current study and review reports of related studies to determine whether the current study needs to be changed or terminated.
  - d) Review proposed modifications to the study prior to their implementation.
  - e) Protect the confidentiality of the accumulated data.
  - f) Determine whether and to whom outcome results should be released prior to the reporting of study results.
  - g) Provide appropriate NIH staff with written information concerning their findings relevant to the quality of the data.

#### References

- 1. Krebs CP, Lindquist CH, Warner TD, Fisher BS, Martin SL. The campus sexual assault study (CSA). Washington, DC: National Institute of Justice, 2007.
- 2. Krebs CP, Lindquist CH, Warner TD, Fisher BS, Martin SL. College women's experiences with physically forced, alcohol- or other drug-enabled, and drug-facilitated sexual assault before and since entering college. J Am Coll Health. 2009;57(6):639-47. Epub 2009/05/13. doi: 10.3200/jach.57.6.639-649. PubMed PMID: 19433402.
- 3. McCauley J, Ruggiero KJ, Resnick HS, Conoscenti LM, Kilpatrick DG. Forcible, drug-facilitated, and incapacitated rape in relation to substance use problems: Results from a national sample of college women. Addictive Behaviors. 2009;34(5):pp. PubMed PMID: Peer Reviewed Journal: 2009-03104-010.
- 4. Senn CY, Eliasziw M, Barata PC, Thurston WE, Newby-Clark IR, Radtke HL, Hobden KL. Sexual violence in the lives of first-year university women in Canada: no improvements in the 21st century. BMC women's health. 2014;14:135. Epub 2014/11/21. doi: 10.1186/s12905-014-0135-4. PubMed PMID: 25410412; PMCID: Pmc4228092.
- 5. DeGue S, Valle LA, Holt MK, Massetti GM, Matjasko JL, Tharp AT. A systematic review of primary prevention strategies for sexual violence perpetration. Aggression and Violent Behavior. 2014;19(4):346-62. doi: http://dx.doi.org/10.1016/j.avb.2014.05.004.
- 6. Salazar LF, VanderEnde K. Date rape prevention in female college students: The last decade in review. Manuscript in preparation. 2015.
- 7. Morrison S, Hardison J, Mathew A, O'Neil J. An evidence-based review of sexual assault preventive intervention programs. Washington, DC: National Instutite of Justice; 2004.
- 8. Gibbons RE. The evaluation of campus-based gender violence prevention programming: What we know about program effectiveness and implications for practitioners. Harrisburg, PA: VAWnet, a project of the National Resource Center on Domestic Violence, 2013.
- 9. Vladutiu CJ, Martin SL, Macy RJ. College- or university-based sexual assault prevention programs: a review of program outcomes, characteristics, and recommendations. Trauma Violence Abuse. 2011;12(2):67-86. Epub 2011/01/05. doi: 10.1177/1524838010390708. PubMed PMID: 21196436.
- 10. Brecklin LR, Forde DR. A meta-analysis of rape education programs. Violence & Victims. 2001;16(3):303-21. PubMed PMID: 11437119.
- 11. Bandura A. Health promotion by social cognitive means. Health Education & Behavior. 2004;31(2):143-64. PubMed PMID: 15090118.
- 12. Abraham C, Michie S. A taxonomy of behavior change techniques used in interventions. Health Psychol. 2008;27(3):379-87. Epub 2008/07/16. doi: 10.1037/0278-6133.27.3.379. PubMed PMID: 18624603.
- 13. Salazar LF, Vivolo-Kantor A, Hardin JW, Berkowitz AD. A Web-based sexual violence bystander intervention for male college students: A randomized controlled trial. Journal of Medical Internet Research. 2014;16(9):e203. doi: 10.2196/jmir.3426.
- 14. Fisher BS, Cullen FT, Turner MG. The sexual vicitimization of college women. In: Justice USDo, editor. Washington: U.S. Department of Justice; 2000.
- 15. Gidycz CA, Dardis CM. Feminist self-defense and resistance training for college students: a critical review and recommendations for the future. Trauma Violence Abuse. 2014;15(4):322-33. Epub 2014/02/06. doi: 10.1177/1524838014521026. PubMed PMID: 24496167.
- 16. Basile KC. A comprehensive approach to sexual violence prevention. New England Journal of Medicine. 2015;372(24):2350-2. doi: doi:10.1056/NEJMe1503952. PubMed PMID: 26061841.
- 17. Banyard VL, Moynihan MM, Plante EG. Sexual violence prevention through bystander education: An experimental evaluation. Journal of Community Psychology. 2007;35(4):463-81.

- 18. Coker AL, Cook-Craig PG, Williams CM, Fisher BS, Clear ER, Garcia LS, Hegge LM. Evaluation of Green Dot: an active bystander intervention to reduce sexual violence on college campuses. Violence against women. 2011;17(6):777-96. Epub 2011/06/07. doi: 10.1177/1077801211410264. PubMed PMID: 21642269.
- 19. Gidycz CA, Orchowski LM, Berkowitz AD. Preventing sexual aggression among college men: An evaluation of a social norms and bystander intervention program. Violence Against Women. 2011;17(6):720-42. doi: 10.1177/1077801211409727. PubMed PMID: 2011-13972-004. First Author & Affiliation: Gidycz, Christine A.
- 20. Gidycz CA, Layman MJ, Rich CL, Crothers M, Gylys J, Matorin A, Jacobs CD. An evaluation of an acquaintance rape prevention program: Impact on attitudes, sexual aggression, and sexual victimization. Journal of Interpersonal Violence. 2001;16(11):1120-38. PubMed PMID: Peer Reviewed Journal: 2001-05182-002.
- 21. Marx BP, Calhoun KS, Wilson AE, Meyerson LA. Sexual revictimization prevention: an outcome evaluation. Journal of Consulting & Clinical Psychology. 2001;69(1):25-32. PubMed PMID: 11302273.
- 22. Senn CY, Eliasziw M, Barata PC, Thurston WE, Newby-Clark IR, Radtke HL, Hobden KL. Efficacy of a sexual assault resistance program for university women. New England Journal of Medicine. 2015;372(24):2326-35. doi: doi:10.1056/NEJMsa1411131. PubMed PMID: 26061837.
- 23. Orchowski LM, Gidycz CA, Raffle H. Evaluation of a sexual assault risk reduction and self-defense program: A prospective analysis of a revised protocol. Psychology of Women Quarterly. 2008;32(2):204-18. PubMed PMID: Peer Reviewed Journal: 2008-05702-009.
- 24. Neilson EC, Gilmore AK, Pinsky HT, Shepard ME, Lewis MA, George WH. The use of drinking and sexual assault protective behavioral strategies: Associations with sexual victimization and revictimization among college women. J Interpers Violence. 2015. Epub 2015/09/09. doi: 10.1177/0886260515603977. PubMed PMID: 26345223.
- 25. Bird ER, Gilmore AK, George WH, Lewis MA. The role of social drinking factors in the relationship between incapacitated sexual assault and drinking before sexual activity. Addict Behav. 2015;52:28-33. Epub 2015/09/09. doi: 10.1016/j.addbeh.2015.08.001. PubMed PMID: 26348279.
- 26. Gilmore AK, Lewis MA, George WH. A randomized controlled trial targeting alcohol use and sexual assault risk among college women at high risk for victimization. Behav Res Ther. 2015;74:38-49. Epub 2015/09/27. doi: 10.1016/j.brat.2015.08.007. PubMed PMID: 26408290.
- 27. Testa M, Parks KA. The role of women's alcohol consumption in sexual victimization. Aggression and Violent Behavior. 1996;1(3):217-34.
- 28. Testa M, Livingston JA. Alcohol consumption and women's vulnerability to sexual victimization: can reducing women's drinking prevent rape? Subst Use Misuse. 2009;44(9-10):1349-76. Epub 2009/11/27. doi: 10.1080/10826080902961468. PubMed PMID: 19938922; PMCID: 2784921.
- 29. Parks KA, Hsieh YP, Bradizza CM, Romosz AM. Factors influencing the temporal relationship between alcohol consumption and experiences with aggression among college women. Psychol Addict Behav. 2008;22(2):210-8. Epub 2008/06/11. doi: 10.1037/0893-164x.22.2.210. PubMed PMID: 18540718; PMCID: 3595014.
- 30. White House Task Force to Protect Students from Sexual Assault. Not Alone: The first report of the White House task force to protect students from sexual assault. Washington, DC: The White House, 2014.
- 31. Nation M, Crusto C, Wandersman A, Kumpfer KL, Seybolt D, Morrissey-Kane E, Davino K. What works in prevention. Principles of effective prevention programs. Am Psychol. 2003;58(6-7):449-56. Epub 2003/09/16. PubMed PMID: 12971191.

- 32. Lewis MA, Neighbors C. Optimizing personalized normative feedback: the use of gender-specific referents. J Stud Alcohol Drugs. 2007;68(2):228-37. Epub 2007/02/09. PubMed PMID: 17286341; PMCID: 2459320.
- 33. Jacobs WJ, Sisco M, Hill D, Malter F, Figueredo AJ. Evaluating theory-based evaluation: information, norms, and adherence. Eval Program Plann. 2012;35(3):354-69. Epub 2012/01/27. doi: 10.1016/j.evalprogplan.2011.12.002. PubMed PMID: 22277114.
- 34. Circle of 6. Circle of 6-WIlliams2015 November 16, 2016. Available from: <a href="http://www.circleof6app.com/downloads/Co6U\_Williams Survey.pdf">http://www.circleof6app.com/downloads/Co6U\_Williams Survey.pdf</a>.
- 35. Salazar LF, DiClemente RJ, Crosby RA. Measurement and design related to theoretically-based health promotion research and practice. Health behavior theory for public health: Principles, foundations and applications. Burlington, MA: Jones & Bartlett Learning; 2013. p. 255-84.
- 36. Crosby RA, Salazar LF, DiClemente RJ. Value expectancy theories. In: DiClemente RJ, Crosby RA, Salazar LF, editors. Health behavior theory for public health: Principles, foundations, and applications. Burlington, MA: Jones & Bartlett Learning; 2013. p. 65-82.
- 37. Noar SM, Zimmerman RS. Health Behavior Theory and cumulative knowledge regarding health behaviors: are we moving in the right direction? Health Education Research. 2005;20(3):275-90. PubMed PMID: 15632099.
- 38. Ashford S, Edmunds J, French DP. What is the best way to change self-efficacy to promote lifestyle and recreational physical activity? A systematic review with meta-analysis. Br J Health Psychol. 2010;15(Pt 2):265-88. Epub 2009/07/10. doi: 10.1348/135910709x461752. PubMed PMID: 19586583.
- 39. Webb TL, Joseph J, Yardley L, Michie S. Using the internet to promote health behavior change: a systematic review and meta-analysis of the impact of theoretical basis, use of behavior change techniques, and mode of delivery on efficacy. J Med Internet Res. 2010;12(1):e4. Epub 2010/02/19. doi: 10.2196/jmir.1376. PubMed PMID: 20164043; PMCID: 2836773.
- 40. Ritterband LM, Thorndike FP, Cox DJ, Kovatchev BP, Gonder-Frederick LA. A behavior change model for internet interventions. Ann Behav Med. 2009;38(1):18-27. Epub 2009/10/06. doi: 10.1007/s12160-009-9133-4. PubMed PMID: 19802647; PMCID: 2878721.
- 41. Hurling R, Fairley BW, Dias MB. Internet-based exercise intervention systems: Are more interactive designs better? Psychology & Health. 2006;21(6):757-72. doi: 10.1080/14768320600603257.
- 42. Salazar LF. Preventing violence against women: A web-based approach. Atlanta, GA: Centers for Disease Control and Prevention; 2013.
- 43. Hust SJ, Marett EG, Lei M, Chang H, Ren C, McNab AL, Adams PM. Health promotion messages in entertainment media: crime drama viewership and intentions to intervene in a sexual assault situation. J Health Commun. 2013;18(1):105-23. Epub 2012/10/02. doi: 10.1080/10810730.2012.688241. PubMed PMID: 23020668.
- 44. Bandura A. Social cognitive theory of mass communication. Bryant, Jennings (Ed); Zillmann, Dolf (Ed). (1994). Media effects: Advances in theory and research. (pp. 61-90); 1994. 505 p.
- 45. Quintero Johnson JM, Harrison K, Quick BL. Understanding the effectiveness of the entertainment-education strategy: an investigation of how audience involvement, message processing, and message design influence health information recall. J Health Commun. 2013;18(2):160-78. Epub 2012/10/04. doi: 10.1080/10810730.2012.688244. PubMed PMID: 23030409.
- 46. Bandura A. Social foundations of thought and action: A social cognitive theory. Englewood Cliffs, NJ: Prentice-Hall; 1986.
- 47. Rozee PD, Koss MP. Rape: A century of resistance. Psychology of Women Quarterly. 2001;25(4):295-311. doi: 10.1111/1471-6402.00030.

- 48. Ullman SE, Knight RA. The efficacy of women's resistance strategies in rape situations. Psychology of Women Quarterly. 1993;17(1):23-38.
- 49. Ullman SE. Review and critique of empirical studies of rape avoidance. Criminal Justice and Behavior. 1997;24(2):177-204.
- 50. Senn CY, Eliasziw M, Barata PC, Thurston WE, Newby-Clark IR, Radtke HL, Hobden KL. Sexual assault resistance education for university women: study protocol for a randomized controlled trial (SARE trial). BMC women's health. 2013;13:25. Epub 2013/05/25. doi: 10.1186/1472-6874-13-25. PubMed PMID: 23702221; PMCID: Pmc3664598.
- 51. Norris J, Nurius PS, Graham TL. When a date changes from fun to dangerous: Factors affecting women's ability to distinguish. Violence against women. 1999;5(3):230-50.
- 52. Nurius PS, Norris J. A Cognitive Ecological Model of Women's Response to Male Sexual Coercion in Dating. Journal of psychology & human sexuality. 1996;8(1-2):117-39. Epub 1996/07/01. doi: 10.1300/J056v08n01 09. PubMed PMID: 25729157; PMCID: Pmc4343209.
- 53. DiClemente RJ, Wingood GM, Harrington KF, Lang DL, Davies SL, Hook EW, 3rd, Oh MK, Crosby RA, Hertzberg VS, Gordon AB, Hardin JW, Parker S, Robillard A. Efficacy of an HIV prevention intervention for African American adolescent girls: a randomized controlled trial. JAMA. 2004;292(2):171-9. PubMed PMID: 15249566.
- 54. Wilson DK, Friend R, Teasley N, Green S, Reaves IL, Sica DA. Motivational versus social cognitive interventions for promoting fruit and vegetable intake and physical activity in African American adolescents. Annals of Behavioral Medicine. 2002;24(4):310-9.
- 55. Orpinas P, Kelder S, Frankowski R, Murray N, Zhang Q, McAlister A. Outcome evaluation of a multi-component violence-prevention program for middle schools: The Students for Peace project. Health Education Research. 2000;15(1):45-58.
- 56. O'Leary A. Social-cognitive theory mediators of behavior change in the National Institute of Mental Health Multisite HIV Prevention Trial. Health Psychology. 2001;20(5):369-76.
- 57. Koniak-Griffin D, Lesser J, Nyamathi A, Uman G, Stein JA, Cumberland WG. Project CHARM: An HIV prevention program for adolescent mothers. Family & Community Health. 2003;26(2):94-107.
- 58. Hallam JS, Petosa R. The long-term impact of a four-session work-site intervention on selected social cognitive theory variables linked to adult exercise adherence. Health Education & Behavior. 2004;31(1):88-100.
- 59. DuRant RH, Barkin S, Krowchuk DP. Evaluation of a peaceful conflict resolution and violence prevention curriculum for sixth-grade students. Journal of Adolescent Health. 2001;28(5):386-93.
- 60. Dilorio C, Resnicow K, Thomas S, Wang DT, Dudley WN, Van Marter DF, Lipana J. Keepin' it R.E.A.L.!: Program description and results of baseline assessment. Health Education & Behavior. 2002;29(1):104-23.
- 61. Anderson ES, Winett RA, Wojcik JR, Winett SG, Bowden T. A computerized social cognitive intervention for nutrition behavior: Direct and mediated effects on fat, fiber, fruits and vegetables, self-efficacy and outcome expectations among food shoppers. Annals of Behavioral Medicine. 2001;23(2):88-100.
- 62. Krueger RA. Focus groups: A practical guide for applied research. 4th ed. Thousand Oaks, CA: Sage Publications, Inc; 2009. 219 p.
- 63. Krueger R, Casey M. Focus groups: A practical guide for applied research. 4th ed. Los Angeles, CA: Sage; 2009. 219 p.
- 64. Clinton-Sherrod M, Morgan-Lopez AA, Brown JM, McMillen BA, Cowell A. Incapacitated sexual violence involving alcohol among college women: the impact of a brief drinking intervention. Violence against women. 2011;17(1):135-54. Epub 2011/01/05. doi: 10.1177/1077801210394272. PubMed PMID: 21199812.
- 65. Cowell AJ, Brown JM, Mills MJ, Bender RH, Wedehase BJ. Cost-effectiveness analysis of motivational interviewing with feedback to reduce drinking among a sample of college

- students. J Stud Alcohol Drugs. 2012;73(2):226-37. Epub 2012/02/16. PubMed PMID: 22333330; PMCID: 3281981.
- 66. Dermen KH, Thomas SN. Randomized controlled trial of brief interventions to reduce college students' drinking and risky sex. Psychol Addict Behav. 2011;25(4):583-94. Epub 2011/09/21. doi: 10.1037/a0025472. PubMed PMID: 21928866; PMCID: 3232340.
- 67. Harris KJ, Catley D, Good GE, Cronk NJ, Harrar S, Williams KB. Motivational interviewing for smoking cessation in college students: a group randomized controlled trial. Prev Med. 2010;51(5):387-93. Epub 2010/09/11. doi: 10.1016/j.ypmed.2010.08.018. PubMed PMID: 20828584; PMCID: 2964425.
- 68. Kazemi DM, Sun L, Nies MA, Dmochowski J, Walford SM. Alcohol screening and brief interventions for college freshmen. J Psychosoc Nurs Ment Health Serv. 2011;49(1):35-42. Epub 2011/01/18. doi: 10.3928/02793695-20101201-02. PubMed PMID: 21235200.
- 69. Martens MP, Smith AE, Murphy JG. The efficacy of single-component brief motivational interventions among at-risk college drinkers. J Consult Clin Psychol. 2013. Epub 2013/03/20. doi: 10.1037/a0032235. PubMed PMID: 23506464.
- 70. Murphy JG, Dennhardt AA, Skidmore JR, Borsari B, Barnett NP, Colby SM, Martens MP. A randomized controlled trial of a behavioral economic supplement to brief motivational interventions for college drinking. J Consult Clin Psychol. 2012;80(5):876-86. Epub 2012/06/06. doi: 10.1037/a0028763. PubMed PMID: 22663899; PMCID: 3435453.
- 71. Murphy JG, Dennhardt AA, Skidmore JR, Martens MP, McDevitt-Murphy ME. Computerized versus motivational interviewing alcohol interventions: impact on discrepancy, motivation, and drinking. Psychol Addict Behav. 2010;24(4):628-39. Epub 2011/01/05. doi: 10.1037/a0021347. PubMed PMID: 21198224.
- 72. Tollison SJ, Mastroleo NR, Mallett KA, Witkiewitz K, Lee CM, Ray AE, Larimer ME. The relationship between baseline drinking status, peer motivational interviewing microskills, and drinking outcomes in a brief alcohol intervention for matriculating college students: a replication. Behav Ther. 2013;44(1):137-51. Epub 2013/01/15. doi: 10.1016/j.beth.2012.09.002. PubMed PMID: 23312433.
- 73. Wagener TL, Leffingwell TR, Mignogna J, Mignogna MR, Weaver CC, Cooney NJ, Claborn KR. Randomized trial comparing computer-delivered and face-to-face personalized feedback interventions for high-risk drinking among college students. J Subst Abuse Treat. 2012;43(2):260-7. Epub 2011/12/27. doi: 10.1016/j.jsat.2011.11.001. PubMed PMID: 22197301.
- 74. Nielsen J. College students on the Web2010 March 15, 2013. Available from: <a href="http://www.nngroup.com/articles/college-students-on-the-web/">http://www.nngroup.com/articles/college-students-on-the-web/</a>.
- 75. Bowen DJ, Kreuter M, Spring B, Cofta-Woerpel L, Linnan L, Weiner D, Bakken S, Kaplan CP, Squiers L, Fabrizio C, Fernandez M. How we design feasibility studies. Am J Prev Med. 2009;36(5):452-7. Epub 2009/04/14. doi: 10.1016/j.amepre.2009.02.002. PubMed PMID: 19362699; PMCID: 2859314.
- 76. Pealer LN, Weiler RM, Pigg RM, Jr., Miller D, Dorman SM. The feasibility of a webbased surveillance system to collect health risk behavior data from college students. Health Educ Behav. 2001;28(5):547-59. Epub 2001/09/29. PubMed PMID: 11575685.
- 77. Baker TB, Brandon TH. Validity of self-reports in basic research. Behavioral Assessment. 1990;12(1):33-51. PubMed PMID: 1990-18701-001.
- 78. Chan D. So why ask me? Are self-report data really that bad? In: Lance CE, Vandenberg RJ, editors. Statistical and methodological myths and urban legends: Doctrine, verity and fable in the organizational and social sciences. New York: Routledge; 2009. p. 309-35.
- 79. James VJ, Lee DR. Through the Looking Glass: Exploring How College Students' Perceptions of the Police Influence Sexual Assault Victimization Reporting. J Interpers Violence. 2014. Epub 2014/10/18. doi: 10.1177/0886260514553116. PubMed PMID: 25324227.

- 80. Gardella JH, Nichols-Hadeed CA, Mastrocinque JM, Stone JT, Coates CA, Sly CJ, Cerulli C. Beyond Clery Act statistics: a closer look at college victimization based on self-report data. J Interpers Violence. 2015;30(4):640-58. Epub 2014/06/14. doi: 10.1177/0886260514535257. PubMed PMID: 24923889.
- 81. Koss MP, Abbey A, Campbell R, Cook S, Norris J, Testa M, Ullman S, West C, White J. Revising the SES: A collaborative process to improve assessment of sexual aggression and victimization. Psychology of Women Quarterly. 2007;31(4):357-70. PubMed PMID: Peer Reviewed Journal: 2007-18440-003.
- 82. Hanson KA, Gidycz CA. Evaluation of a sexual assault prevention program. Journal of Consulting & Clinical Psychology. 1993;61(6):1046-52. PubMed PMID: 8113482.
- 83. Breitenbecher KH. The convergent validities of two measures of dating behaviors related to risk for sexual victimization. J Interpers Violence. 2008;23(8):1095-107. Epub 2008/02/15. doi: 10.1177/0886260507313974. PubMed PMID: 18272726.
- 84. Moore CD, Waterman CK. Predicting self-protection against sexual assault in dating relationships among heterosexual men and women, gay men, lesbians, and bisexuals. Journal of College Student Development. 1999;40(2):132-40. PubMed PMID: Peer Reviewed Journal: 1999-10727-002.
- 85. Martens MP, Ferrier AG, Sheehy MJ, Corbett K, Anderson DA, Simmons A. Development of the protective behavioral strategies survey. J Stud Alcohol. 2005;66(5):698-705. Epub 2005/12/07. PubMed PMID: 16329461.
- 86. Collins JJ, Messerschmidt PM. Epidemiology of alcohol-related violence. Alcohol Health and Research World. 1993;17(2):93-100.
- 87. Tyler KA, Schmitz RM, Adams SA. Alcohol expectancy, drinking behavior, and sexual victimization among female and male college students. J Interpers Violence. 2015. Epub 2015/07/02. doi: 10.1177/0886260515591280. PubMed PMID: 26130688.
- 88. George WH, Frone MR, Cooper ML, Russell M, Skinner JB, Windle M. A revised Alcohol Expectancy Questionnaire: factor structure confirmation, and invariance in a general population sample. Journal of Studies on Alcohol. 1995;56(2):177-85.
- 89. Baer JS, Stacy A, Larimer M. Biases in the perception of drinking norms among college students. J Stud Alcohol. 1991;52(6):580-6. Epub 1991/11/01. PubMed PMID: 1758185.
- 90. Dietz S, Blackwell KT, Daley PC, Bentley BJ. Measurement of empathy toward rape victims and rapists. Journal of Personality and Social Psychology. 1982;43:372-84.
- 91. Dilorio C, Parsons M, Lehr S, Adame D, Carlone J. The psychometric evaluation of an instrument to measure safe sex behaviors in adolescents and young adults. Nursing Research. 1992;41:203-6.
- 92. Dilorio C, Dudley WN, Lehr S, Soet JE. Correlates of safer sex communication among college students. Journal of Advanced Nursing. 2000;32(3):658-65.
- 93. Ozer EM, Bandura A. Mechanisms governing empowerment effects: a self-efficacy analysis. Journal of Personality & Social Psychology. 1990;58(3):472-86. PubMed PMID: 2324938.
- 94. Binik YM, Mah K, Kiesler S. Ethical issues in conducting sex research on the Internet. The Journal of Sex Research. 1999;36(1):82-90.
- 95. Schulz KF, Altman DG, Moher D. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. BMC medicine. 2010;8(1):18.
- 96. Stephenson R Fau Rentsch C, Rentsch C Fau Salazar LF, Salazar Lf Fau Sullivan PS, PS S. Dyadic Characteristics and Intimate Partner Violence among Men Who Have Sex with Men. West J Emerg Med. 2011;12(3):324-32.
- 97. Salazar LF, Stephenson RB, Sullivan PS, Tarver R. Development and validation of HIV-related dyadic measures for men who have sex with men. J Sex Res. 2013;50(2):164-77. Epub 2011/12/31. doi: 10.1080/00224499.2011.636845. PubMed PMID: 22206480.

- 98. Cameron KA, Salazar LF, Bernhardt JM, Burgess-Whitman N, Wingood GM, DiClemente RJ. Adolescents' experience with sex on the web: Results from online focus groups. Journal of Adolescence. 2005;28(4):535-40.
- 99. Sullivan PS, Peterson J, Rosenberg ES, Kelley CF, Cooper H, Vaughan A, Salazar LF, Frew P, Wingood G, Diclemente R, del Rio C, Mulligan M, Sanchez TH. Understanding racial HIV/STI disparities in black and white men who have sex with men: a multilevel approach. PLOS one. 2014;9(3):e90514. Epub 2014/03/13. doi: 10.1371/journal.pone.0090514. PubMed PMID: 24608176; PMCID: 3946498.
- 100. Hennessy M, Romer D, Valois RF, Vanable P, Carey MP, Stanton B, Brown L, DiClemente R, Salazar LF. Safer sex media messages and adolescent sexual behavior: 3-year follow-up results from project iMPPACS. Am J Public Health. 2013;103(1):134-40. Epub 2012/11/17. doi: 10.2105/ajph.2012.300856. PubMed PMID: 23153149; PMCID: Pmc3518371.
- 101. Diggle PJ, Heagerty P, Liang KY, Zeger SL. Analysis of longitudinal data. Oxford, U.K.: Clarendon Press; 2002.
- 102. Preacher KJ, Hayes AF. SPSS and SAS procedures for estimating indirect effects in simple mediation models. Behavior Research Methods, Instruments, & Computers. 2004;36(4):717-31.
- 103. MacKinnon DP, Lockwood CM, Hoffman JM, West SG, Sheets V. A comparison of methods to test mediation and other intervening variable effects. Psychological methods. 2002;7(1):83-104.
- 104. Testa M, Hoffman JH, Livingston JA, Turrisi R. Preventing college women's sexual victimization through parent based intervention: a randomized controlled trial. Prev Sci. 2010;11(3):308-18. Epub 2010/02/20. doi: 10.1007/s11121-010-0168-3. PubMed PMID: 20169410; PMCID: 2904876.
- 105. Testa M, VanZile-Tamsen C, Livingston JA, Koss MP. Assessing women's experiences of sexual aggression using the Sexual Experiences Survey: Evidence for validity and implications for research. Psychology of Women Quarterly. 2004;28(3):256-65.
- 106. Livingston JA, Testa M, VanZile-Tamsen C. The reciprocal relationship between sexual victimization and sexual assertiveness. Violence against women. 2007;13(3):298-313.
- 107. Testa M, Hoffman JH, Livingston JA. Alcohol and sexual risk behaviors as mediators of the sexual victimization–revictimization relationship. Journal of consulting and clinical psychology. 2010;78(2):249.
- 108. Kypri K, Saunders JB, Gallagher SJ. Acceptability of various brief intervention approaches for hazardous drinking among university students. Alcohol & Alcoholism. 2003;38(6):626-8.
- 109. Neighbors C, Larimer ME, Lewis MA. Targeting misperceptions of descriptive drinking norms: Efficacy of a computer-delivered personalized normative feedback intervention. Journal of Consulting and Clinical Psychology. 2004;72(3):434-47. PubMed PMID: Peer Reviewed Journal: 2004-95166-007.
- 110. Khadaroo ST. UConn setlles sexual assault suit for \$1.2 million. Will more schools be sued? The Christian Science Monitor [Internet]. 2014. Available from: <a href="http://www.csmonitor.com/USA/Education/2014/0718/UConn-settles-sexual-assault-suit-for-1.2-million.-Will-more-schools-be-sued-video">http://www.csmonitor.com/USA/Education/2014/0718/UConn-settles-sexual-assault-suit-for-1.2-million.-Will-more-schools-be-sued-video</a>.
- 111. Anderson N. Tally of federal probes of colleges on sexual violence grows 50 percent since may. The Washington Post [Internet]. 2014 November 12, 2014. Available from: <a href="http://www.washingtonpost.com/local/education/tally-of-federal-probes-of-colleges-on-sexual-violence-grows-50-percent-since-may/2014/10/19/b253f02e-54aa-11e4-809b-8cc0a295c773\_story.html">http://www.washingtonpost.com/local/education/tally-of-federal-probes-of-colleges-on-sexual-violence-grows-50-percent-since-may/2014/10/19/b253f02e-54aa-11e4-809b-8cc0a295c773\_story.html</a>.
- 112. White House Council on Women and Girls and the Office of the Vice President. Rape and sexual assault: A renewed call to action. Washington, DC: The White House, 2014.